CLINICAL TRIAL: NCT07358520
Title: Prospective, Multicenter, Parallel-Controlled Clinical Study on the Use of Huaier Granules for the Treatment of Bevacizumab- and Anlotinib-Related Proteinuria in Lung Cancer Patients
Brief Title: Clinical Study on the Use of Huaier Granules for the Treatment of Proteinuria Related to Bevacizumab and Anlotinib in Lung Cancer Patients
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Jialei Wang, Professor, Fudan University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HE-202508
Record Dates: First submitted 2026-01-14; First posted 2026-01-22 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Proteinuria
Keywords: Huaier Granules; Proteinuria; Bevacizumab; Anlotinib
MeSH Terms: conditions — Proteinuria | interventions — anlotinib; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Huaier Granules (Experimental): Take orally, 10g each time, three times a day. Participants in the experimental group should continue treatment for at least 24 weeks or until treatment failure, intolerable toxicity, withdrawal from the study for any reason, or death, whichever occurs first; or until the investigator determines that there is no further benefit. For specific usage, refer to the drug instructions.
  Interventions: Drug: Huaier Granule
- Anlotinib and Bevacizumab (Active Comparator): Administer according to clinical routine practice. Refer to the respective drug prescribing information for specific usage. Continue treatment until disease progression, intolerable toxicity, withdrawal from the study for any reason, or death, whichever occurs first.
  Interventions: Drug: Anlotinib and Bevacizumab

INTERVENTIONS:
Drug: Huaier Granule — Take orally, 10g each time, three times daily.
  Arms: Huaier Granules
Drug: Anlotinib and Bevacizumab — Administer according to clinical routine practice. Refer to the respective drug prescribing information for specific usage.
  Arms: Anlotinib and Bevacizumab

SUMMARY:
This study is a prospective, multicenter, parallel-controlled clinical trial designed to evaluate the therapeutic efficacy of Huaier Granules for proteinuria occurring in lung cancer patients undergoing treatment with either Bevacizumab or Anlotinib.

DETAILED DESCRIPTION:
This study is a prospective, multicenter, parallel-controlled exploratory trial. It plans to enroll 40 subjects diagnosed with malignant lung tumors, who will visit the selected research centers from October 2025 to October 2026. All subjects will be assigned to either the control group or the experimental group based on clinical management and their own preference. Subjects in the control group will receive no therapeutic intervention, while those in the experimental group will be administered Huaier Granules.Throughout the study period, the planned duration for subject recruitment and enrollment is 12 months. The total follow-up duration for enrolled subjects is 48 weeks. After enrollment, subjects will be followed up every 2 weeks during the first 8 weeks, and then every 4 weeks thereafter. Follow-ups will continue until the study ends, the subject withdraws from the study for any reason, is lost to follow-up, or dies, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years;
* Histopathologically confirmed diagnosis of lung cancer;
* Receiving Bevacizumab or Anlotinib treatment;
* Positive urine protein detection, with 0.15g < 24-hour urinary protein quantification < 3.5g;
* No treatment with Huaier Granules within one month prior to enrollment;
* Expected survival time not less than 6 months;
* Voluntary participation in this study and provision of signed informed consent.

Exclusion Criteria:

* Known allergy, contraindication, or caution to any component of Huaier Granules;
* Inability to take oral medication;
* Required or ongoing use of drugs known to potentially affect proteinuria, including but not limited to ACE inhibitors, glucocorticoids (>3 weeks), and Chinese patent medicines (as per respective drug prescribing information);
* Proteinuria caused by underlying diseases, including but not limited to nephropathy, hypertension, urinary tract infection, systemic lupus erythematosus, multiple myeloma, etc.;
* Women who are pregnant, breastfeeding, or planning pregnancy;
* Currently participating in other clinical trials investigating drugs for treating proteinuria;
* Refusal to cooperate with follow-up;
* Any other reasons deemed by the investigator as unsuitable for participation in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2026-01-28 (Estimated); Primary Completion 2027-01-28 (Estimated); Study Completion 2028-01-28 (Estimated)

PRIMARY OUTCOMES:
16-week Efficacy Rate for Proteinuria Treatment | Start of treatment until 16-week follow-up
  It defined as the proportion of subjects achieving complete remission, partial remission, or stable disease according to proteinuria treatment efficacy evaluation at 16 weeks, relative to the total number of subjects in both groups.

SECONDARY OUTCOMES:
48-week Recurrence Rate for Proteinuria Treatment | Start of treatment until 48-week follow-up
  It defined as the proportion of subjects whose proteinuria reverts to positive (≥1+) after becoming negative during treatment, relative to the total number of subjects.
48-week Resumption and Discontinuation Rates for Bevacizumab or Anlotinib after Proteinuria Treatment | Start of treatment until 48-week follow-up
  It defined as the proportion of subjects who, due to worsening proteinuria, required temporary suspension of bevacizumab or anlotinib and subsequently resumed treatment after proteinuria alleviation, relative to the total number of subjects.
Incidence and Severity of Other Adverse Reactions (including but not limited to hypertension, bleeding, and gastrointestinal perforation) after 48 weeks of Proteinuria Treatment | Start of treatment until 48-week follow-up
  Incidence is defined as the proportion of subjects experiencing other adverse reactions (including but not limited to hypertension, bleeding, and gastrointestinal perforation) relative to the corresponding total population. Severity will be assessed as per the relevant descriptions in the adverse event definitions and evaluation section

CONTACTS AND LOCATIONS:
Overall Officials: Jialei Wang, phD, Principal Investigator — Fudan University
Locations (2):
- China (2):
  - Xuzhou Central Hospital, Xuzhou, Jiangsu
  - Xin Hua Hospital Affiliated to Shanghai Jiao Tong University School of Medicine, Shanghai, Shanghai Municipality

IPD SHARING:
Plan to Share IPD: No